CLINICAL TRIAL: NCT05705622
Title: The Effect of Nursing Education on Oral Mucositis in Bone Marrow Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Collaborators: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Recep Turan, Medical Nurse, MSc, Antalya Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2010
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Blood Stem Cell Transplant Failure; Oral Mucositis; Nurse's Role
Keywords: Blood Stem Cell Transplantation; Oral Mucositis; Nurse Education for Patients
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial. Oral mucositis levels of patients treated in hospital for bone marrow transplantation will be examined. Before starting the research, permission will be obtained from the patients, and after the necessary randomization, they will be assigned to the experimental and control groups. The patients in the experimental group will be trained for oral mucositis. Oral diagnosis of the patients will be made once a week for four weeks and the effectiveness of the nursing education given to the patients will be evaluated.
Who Masked: Participant
Masking Description: This study will be conducted by a researcher. Patients will be assigned to the experimental and control groups after the randomization process. Patients will not know which group they are in. In this study, only the researcher will know which group the patients are in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental intervention group (Experimental): Sociodemographic information, comorbidity, habits and disease information of the patients included in the experimental group were obtained through the Patient Diagnosis Form and recorded in the form. The patients were evaluated for oral mucositis by diagnosing the mouth. It was recorded in the World Health Organization Mucositis Evaluation Form, Oral Mucositis Risk Assessment Scale in Hematology Patients, Oral Mucous Membrane Evaluation and Follow-up Form. After the diagnosis of oral mucositis was made, a pre-test was performed using the "Oral Mucositis Knowledge Level Evaluation Form" to measure the oral mucositis knowledge level of the patients. Later, the patients included in the experimental group were given training on the evaluation, prevention, care and treatment of oral mucositis, and a training booklet was given for the benefit of the patients.
  Interventions: Other: Oral mukositis nurse's education for patients
- No intervention control group (No Intervention): The first follow-up of the patients included in the control group was made in the patient's room on the day of their admission to the bone marrow transplant unit. Sociodemographic information, comorbidity, habits and disease information of the patients were obtained through the Patient Diagnosis Form and recorded in the form. The patients were evaluated for oral mucositis by diagnosing the mouth. It was recorded in the World Health Organization Mucositis Evaluation Form, Oral Mucositis Risk Assessment Scale in Hematology Patients, Oral Mucous Membrane Evaluation and Follow-up Form. The patients in the control group were not given training on oral mucositis and the training booklet prepared by the researcher was not given.

INTERVENTIONS:
Other: Oral mukositis nurse's education for patients — Education given to patients by nurses on the prevention, treatment and care of oral mucositis
  Arms: Experimental intervention group

SUMMARY:
In this study, it is aimed to examine the effect of oral care training for oral mucositis, which will be given by the researcher to patients who have undergone bone marrow transplantation, on the incidence and severity of oral mucositis in patients. The aim of the study is to be carried out in a public and private hospital in Antalya province, in two different hospitals with a public and private status, and with a total of 60 patients, 30 of which are in the experimental group and 30 in the control group. In the study, "oral care training for oral mucositis" and "oral mucositis follow-up procedure" will be developed by the researcher for bone marrow transplant patients. Bone marrow transplant patients will be educated and followed up according to the follow-up procedure before starting the chemotherapy regimen treatments planned before the transplant.

DETAILED DESCRIPTION:
Type of study: It was designed as a randomized controlled experimental study.

Location and Characteristics of the Research:

With the application for the Permission of the Research Ethics Committee, the official institution permission process was started and the Medstar Antalya Hospital was approved by Prof. Dr. It is planned to be performed in İhsan Karadoğan Bone Marrow Transplantation unit and in the Adult Bone Marrow Transplantation Unit of Akdeniz University Medical Faculty Hospital. prof. Dr. İhsan Karadoğan bone marrow transplant unit has a total of 19 beds and 16 KIT nurses work. There are 12 patient beds and 11 KIT nurses work in the Adult Bone Marrow Transplant Unit of Akdeniz University Medical Faculty Hospital. In both units, the rooms have a positive pressure system, air filtration is provided with the hepafilter system, it works with private rooms and a system of having only one attendant.

Population and Sample of the Research:

The population of the study will consist of individuals over 17 years of age, who are hospitalized in the relevant clinics and have been decided to have a bone marrow transplant, who can speak Turkish and who have no communication barriers, who are prepared for transplantation, and who do not have oral mucositis in their mouths. The research sample will consist of patients who have these characteristics and agree to participate in the study. Patients will be randomly assigned to the experimental and control groups.

The targeted situation with this study; The aim of the study is to reduce the development of intraoral infections due to the decrease of immune resistance of the patients after the transplantation with the effect of the chemotherapy treatment given before the transfer of the nurse training given for oral mucositis or the degree of the developing oral mucositis, the severity of the pain, its effect on nutrition, speech and swallowing power. Another goal of this study is to enable patients to know the effects of oral mucositis that may develop during the transplant process and to manage this process effectively.

Analysis of Data:

The analysis of the obtained data will be evaluated with SPSS 20.0 package programs. The normal distribution of the data will be checked with the Shapiro-Wilk test. Independent two-sample t-test will be used to compare normally distributed data, and Manny-Whitney U-test will be used for non-normally distributed data. In the comparison of the pre-test and post-test data of the experimental (educational) and control groups, dependent sample t-test will be used for normally distributed variables, and Wilcoxon t-test will be used for non-normally distributed variables. Chi-square (X2) test exact values will be used in the comparison of categorical variables. The relationships of continuous data will be looked at with Spearman's rho correlation analysis. Statistical significance level will be accepted as p<0.05 in all analyzes.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 17 who will undergo bone marrow transplantation
* Patients who can speak Turkish and have no communication barriers
* Patients without oral mucositis during preparation for bone marrow transplant

Exclusion Criteria:

* Under 18 years old
* Patients who do not speak Turkish and have communication barriers
* Patients with oral mucositis during bone marrow transplant preparation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Patient Diagnosis Form | 4 months
  include 16 ask about diagnosis of patients
Mucositis Evaluation Form of the World Health Organization | 4 months
  WHO mucositis scores 0 (no symptoms), 1 (oral pain) erythema - no change in oral intake, 2 (oral erythema and ulcers, strict diet tolerated - soft foods only), 3 (oral ulcers, liquid diet only) and 4 ( oral feeding is impossible). High scores for the WHO mucositis scale indicate severe mucositis.
Oral Mucositis Risk Assessment Scale in Hematology Patients | 3 months
  The duration of evaluating the risk of developing OM in hematology patients consisted of a total of 11 items. The cut-off point of the scale was found to be 11.5. However, the use of 12 points as the cut-off point in clinical use, and the patients who score 12 points or more are those who have the risk of developing OM.
Oral Mucous Membrane Evaluation and Follow-up Form | 2 months
  Each category is evaluated by talking to the patient, observing the oral cavity, and using the hand or spatula, and 1 point if normal, 2 points if cracked voice, pain during swallowing, dry or chapped lips, redness, dark or sticky saliva, difficulty speaking or if there is pain, inability to swallow, ulceration or bleeding, 3 points are given. The total score of the guide varies between 8 and 24. An increase in score indicates an increased risk of developing mucositis or occurrence of mucositis, taking into account the changed parameters.
Oral Mucous Membrane Evaluation and Follow-up Form | 1 months
  It consists of 20 questions covering oral mucositis treatment, oral care and oral mucositis management.

CONTACTS AND LOCATIONS:
Overall Officials: Kamuran Cerit, Study Director — Antalya Training Research and Hospital
Locations (1):
- Süleyman Demirel Üniversitesi, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: World Health Organization. WHO handbook for reporting results of cancer treatment. — https://apps.who.int/iris/handle/10665/37200